CLINICAL TRIAL: NCT03904043
Title: Non-Operative Management and Early Response Assessment in Rectal Cancer
Acronym: NOM-ERA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201904029
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Adenocarcinoma of the Lower Rectum
MeSH Terms: interventions — Radiotherapy; Folfox protocol; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Radiation + FOLFOX (Experimental): * Pelvic radiotherapy 5GY x 5 fractions once daily
  * Radiation to extra-mesorectal node 7 Gy x 5 fractions once daily
  * FOLFOX should begin 2-4 weeks after completion of radiotherapy and will consist of FOLFOX x 8 cycles (16 weeks).
    * Oxaliplatin day 1 every 14 days
    * Leucovorin day 1 every 14 days. Levoleucovorin may be substituted if leucovorin is not available.
    * 5-FU bolus day 1 every 14 days
    * 5-FU infusion day 1 every 14 days over 46 hours
  * An optional simultaneous integrated boost of 30 Gy in 5 fractions to the primary tumor is permitted
  Interventions: Radiation: Radiation therapy; Drug: FOLFOX regimen
- Radiation + CAPOX (Experimental): * Pelvic radiotherapy 5GY x 5 fractions once daily
  * Radiation to extra-mesorectal node 7 Gy x 5 fractions once daily
  * CAPOX should begin 2-4 weeks after completion of radiotherapy and will consist of CAPOX x 5 cycles (15 weeks).
    * Capecitabine 1000 mg/m^2 by mouth twice per day on days 1-14 of every 21 day cycle
    * Oxaliplatin 130 mg/m^2 intravenous on day 1 of each 21 day cycle
  * An optional simultaneous integrated boost of 30 Gy in 5 fractions to the primary tumor is permitted
  Interventions: Radiation: Radiation therapy; Drug: CAPOX regimen

INTERVENTIONS:
Radiation: Radiation therapy — -Monday-Friday treatment is strongly recommended
Drug: FOLFOX regimen — -CAPOX can be given as alternative
  Arms: Radiation + FOLFOX
Drug: CAPOX regimen — Given as an alternative to FOLFOX
  Arms: Radiation + CAPOX

SUMMARY:
The investigators' data from a phase I study of short course radiation therapy followed by chemotherapy showed 74% complete clinical response (cCR). Given the promising response rate, the investigators are evaluating short course radiation therapy (SCRT) followed by chemotherapy in a multi-institution phase II trial to validate the cCR rate of this treatment paradigm. SCRT has not been prospectively evaluated in non-operative management for patients with non-metastatic rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biopsy proven stage I-IIIB (cT1-3, N0-2a, M0) adenocarcinoma of the rectum; staging must also be based on multidisciplinary evaluation including MRI
* Tumor ≤ 12 cm from anal verge as determined by MRI or endoscopy
* Clinically detectable (MR, endoscopy, or DRE) tumor present
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least 18 years of age
* Adequate bone marrow function defined as:

  * Absolute neutrophil count (ANC) > 1,500 cells/mm3
  * Hemoglobin> 8 g/dl
  * Platelets >100,000 cells/mm3
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent document.

Exclusion Criteria

* Prior radiation therapy, chemotherapy or extirpative surgery for rectal cancer.
* Prior oxaliplatin or capecitabine use for any malignancy
* No prior radiation therapy to the pelvis.
* A history of other malignancy (except non-melanomatous skin cancers) with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Currently receiving any investigational agents.
* A history of allergic reaction attributed to compounds of similar chemical or biologic composition to capecitabine, 5FU, oxaliplatin, or leucovorin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective antiretroviral therapy (ART) according to Department of Health and Human Services (DHHS) treatment guidelines is recommended. HIV testing for patients without a history of HIV is not a protocol requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Waters, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with investigators who submit a sound proposal. Participants who opted out of data sharing in the informed consent will not be included.
Time Frame: Up to 5 years after completion of the study
Access Criteria: Proposals should be directed to kim.hyun@wustl.edu. To gain access, data requestors will need to sign a data access agreement and provide proof of appropriate regulatory approvals as necessary.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation + FOLFOX | Radiation + CAPOX
Started | 55 | 8
Completed | 51 | 7
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Did not start treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation + FOLFOX | Radiation + CAPOX | Total
Number analyzed (Participants) | 55 | 8 | 63
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 84] | 60 [34 to 72] | 61 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 2 | 19
  Male | 38 | 6 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 55 | 8 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 49 | 7 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 8 | 63

OUTCOME MEASURES:

1. Primary Outcome: Clinical Complete Response Rate
Description: - Criteria for clinical complete response:
  * No residual gross tumor at procto/sigmoidoscopy; or only erythematous scar or ulcer
  * No palpable tumor on DRE
  * No radiographic evidence of tumor on MRI
  * No suspicious mesorectal lymph nodes on MRI
  * Negative biopsy from scar, ulcer, or former tumor site (if necessary according to surgeon's judgment)
Time Frame: Completion of treatment (estimated to be 22 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + FOLFOX | Radiation + CAPOX
Number analyzed (Participants) | 51 | 7
Participants | 36 | 2

2. Secondary Outcome: Progression-free Survival (PFS)
Description: * Criteria for progressive disease:
    * Increase in the size of primary tumor by RECIST criteria (increase of at least 20% from nadir in the sum of the target lesion, with an absolute increase of at least 5 mm)
    * New metastatic disease
  * PFS is defined as the time from date of treatment to death or progression, which occurs first. The alive patients without progression are censored as the last date follow-up.
Time Frame: At 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Any Grade 3 or Higher Toxicity During Treatment
Description: - The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: From start of treatment through the completion of treatment (estimated to be 22 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation + FOLFOX | Radiation + CAPOX
Number analyzed (Participants) | 54 | 8
Participants
  Abdominal pain | 0 | 1
  Acidosis | 1 | 0
  Alanine aminotransferase increased | 2 | 0
  Anal pain | 0 | 1
  Anemia | 1 | 1
  Anorexia | 0 | 2
  Anxiety | 0 | 1
  Aspartate aminotransferase increased | 1 | 0
  Congestive heart failure | 1 | 0
  Dehydration | 1 | 0
  Delirium | 0 | 1
  Depression | 0 | 1
  Diarrhea | 5 | 1
  Fall | 1 | 1
  Fatigue | 1 | 1
  Febrile neutropenia | 1 | 0
  Generalized muscle weakness | 1 | 1
  Hyperglycemia | 3 | 0
  Hypertension | 1 | 0
  Hypoalbuminemia | 0 | 1
  Hypocalcemia | 0 | 1
  Hypokalemia | 2 | 0
  Hyponatremia | 1 | 0
  Infection - cellulitis | 1 | 0
  Neutrophil count decreased | 22 | 1
  Peripheral sensory neuropathy | 1 | 1
  Platelet count decreased | 0 | 1
  Proctitis | 2 | 1
  Rectal hemorrhage | 1 | 0
  Rectal pain | 0 | 1
  Skin infection | 1 | 0
  Superior vena cava syndrome | 1 | 0
  Thromboembolic event | 1 | 1
  Vomiting | 0 | 1
  Weight loss | 0 | 1
  White blood cell decreased | 7 | 0

4. Secondary Outcome: Incidence of Post Chemoradiotherapy Grade 3 or Higher Toxicity
Description: as for outcome 3
Time Frame: At 1 year after the start of radiation
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Anorectal Function as Measured by the FACT-C Questionnaire
Description: * Questionnaire with 5 sections (physical well-being, social/family well being, emotional well-being, functional well-being, and additional concerns)
  * Answers to the questions range from 0=not at all to 4=very much. The higher the total score the lower quality of life.
Time Frame: 10-14 months after radiation therapy
Reporting Status: Not Posted

6. Secondary Outcome: Organ Preservation Rate
Time Frame: At 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Organ Preservation Rate
Time Frame: At 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 1 year after the start of radiation therapy. All-cause mortality was collected from start of treatment through completion of follow-up (up to 2 years after completion of chemoradiation).
Description: Grade 1-2 adverse events were not collected per protocol unless they were considered a serious adverse event.
Arm/Group | Radiation + FOLFOX | Radiation + CAPOX
All-Cause Mortality (participants affected / at risk) | 1/54 | 0/8
Serious Adverse Events (participants affected / at risk) | 21/54 | 2/8
Other Adverse Events (participants affected / at risk) | 28/54 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation + FOLFOX (N=54) | Radiation + CAPOX (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Intestinal malrotation (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Hematoma (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Idiopathic hypotension (Injury, poisoning and procedural complications) | 1 | 0
Ileostomy complications (Injury, poisoning and procedural complications) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Hydroephrosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation + FOLFOX (N=54) | Radiation + CAPOX (N=8)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Congestive heart failure (Cardiac disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1
Proctitis (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 0
Neutrophil count decreased (Investigations) | 17 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 6 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03904043/Prot_SAP_001.pdf